CLINICAL TRIAL: NCT01599741
Title: Clinical Validation and Evaluation of X-ray Image Processing for Endovascular Digital Subtraction Angiography and Intervention
Brief Title: X-ray Dose Reduction Study for Endovascular Interventional Radiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: XCY607-100093
Record Dates: First submitted 2012-05-08; First posted 2012-05-16 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Disease
Keywords: X-rays; Endovascular angiography; Image processing
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ClarityIQ (Experimental): Low-dose DSA (83% reducation compared to normal dose) with novel X-ray imaging technology.
  Interventions: Radiation: Low-dose DSA (83% reduction compared to normal dose) with novel X-ray imaging technology.
- AlluraXper (Active Comparator): Normal dose DSA with conventional X-ray imaging technology.
  Interventions: Radiation: Normal dose DSA with conventional X-ray imaging technology

INTERVENTIONS:
Radiation: Low-dose DSA (83% reduction compared to normal dose) with novel X-ray imaging technology. — Digital Subtraction Angiography (DSA) of iliac artery with reduced dose settings (83% dose reduction expected) in combination with novel X-ray imaging technology.
  Other Names: ClarityIQ
  Arms: ClarityIQ
Radiation: Normal dose DSA with conventional X-ray imaging technology — Digital Subtraction Angiography (DSA) of iliac artery with normal dose settings in combination with conventional X-ray imaging technology.
  Other Names: AlluraXper
  Arms: AlluraXper

SUMMARY:
ClarityIQ is a novel X-ray imaging technology, that combines advanced real-time image noise reduction algorithms, with state-of-the-art hardware to reduce patient entrance dose significantly. This is realized by anatomy-specific optimization of the full acquisition chain (grid switch, beam filtering, pulse width, spot size, detector and image processing engine) for every clinical task individually. Furthermore, smaller focal spot sizes, shorter pulses and the introduction of automatic real-time motion compensation in subtraction imaging are used, which are known to positively influence image quality . The final effect on the clinical image quality in peripheral angiography is investigated in this study.

DETAILED DESCRIPTION:
X-ray dose and image quality are related by laws of physics. Low dose and high image quality cannot be achieved at the same time. However, image processing algorithms can help an x-ray system to acquire images with lower dose without influencing image quality or achieving higher image quality with equal dose. The primary aim of this study is to verify if the diagnostic image quality is equal or better when using a significant reduction in X-ray dose for endovascular digital subtraction angiography in combination with a novel imaging technology compared to using normal dose with conventional image technology.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age undergoing digital subtraction angiography for diagnosis or treatment of iliac artery disease.

Exclusion Criteria:

* Patients not willing or unable to give consent to participate
* Patients already involved in a clinical trial
* Patients under the age of 18
* Pregnant or breastfeeding women
* Patients with kidney disease (eGFR < 60)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco van Strijen, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of patients occured between July 3 and October 12, 2012
Groups:
- Allura-Xper-ClarityIQ: DSA acquisition of iliac artery with AlluraXper directly followed by DSA with ClarityIQ
Period: Overall Study
Arm/Group | Allura-Xper-ClarityIQ
Started | 51
Collected Dose and Image Information | 48
Completed | 48
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Allura-Xper-ClarityIQ: DSA acquisition of iliac artery with AlluraXper followed by DSA with ClarityIQ
Arm/Group | Allura-Xper-ClarityIQ
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 35
Region of Enrollment [Number; unit: participants]
  Netherlands | 51

OUTCOME MEASURES:

1. Primary Outcome: Image Quality
Description: Overall proportion where diagnostic image quality of ClarityIQ is scored equal or better compared to AlluraXper by the blinded reviewers. Reading is performed by simultaneous visual comparison of image quality of AlluraXper and ClarityIQ by multiple blinded readers. All blinded readers have rated all side-by-side presented images. The images are presented in a random order and blinded to the reader. The hypothesis is that the overall proportion where diagnostic image quality of ClarityIQ is scored equal or better is ≥ than 0.80. Combined for all raters, the lower bound of the one-sided 95% CI (lower bound of the two-sided 90% CI) is used.
Time Frame: 1 Day
Population: All patients with recorded dose information from the system for both DSA runs were used.
Measure: Mean (90% Confidence Interval); unit: Proportion of images rated equal/better
Groups:
- Allura-Xper-ClarityIQ: DSA acquisition of iliac artery with AlluraXper followed by DSA with ClarityIQ or visa versa.
Arm/Group | Allura-Xper-ClarityIQ
Number analyzed (Participants) | 48
Proportion of images rated equal/better | 0.96 [0.93 to 0.98]

2. Secondary Outcome: Radiation Dose Measurements: Dose Area Product (DAP)
Description: Percentage dose change of ClarityIQ vs. AlluraXper in DAP calculated by DAP/frame for DSA. Negative change means a reduction in dose for ClarityIQ vs. AlluraXper.
  DAP was measured during the ClarityIQ and AlluraXper runs during the procedure.
Time Frame: Participants were followed for the duration of the procedure
Population: All patients with recorded dose information from the system for both DSA runs were used.
Measure: Mean (Standard Deviation); unit: percentage of dose change
Arm/Group | Allura-Xper-ClarityIQ
Number analyzed (Participants) | 48
percentage of dose change | -83 (5)

3. Secondary Outcome: Radiation Dose Measurements: Air Kerma (AK)
Description: Percentage dose change of ClarityIQ vs. AlluraXper in AK calculated by AK/frame for DSA. Negative change means a reduction in dose for ClarityIQ vs. AlluraXper.
  AK was measured during the ClarityIQ and AlluraXper runs during the procedure.
Time Frame: Participants were followed for the duration of the procedure
Population: All patients with recorded dose information from the system for both DSA runs were used.
Measure: Mean (Standard Deviation); unit: percentage of dose change
Arm/Group | Allura-Xper-ClarityIQ
Number analyzed (Participants) | 48
percentage of dose change | -83 (5)

ADVERSE EVENTS:
Time Frame: Procedure
Arm/Group | Allura-Xper-ClarityIQ
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less